CLINICAL TRIAL: NCT03301428
Title: Effectiveness of Different Educational Tools to Improve Beliefs About Pain and Reduce Pain-related Disability in Patients With Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Educational Tools to Improve Beliefs About Pain and Reduce Pain-related Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Christophe Demoulin, Invited Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLBP EDUC
Record Dates: First submitted 2017-09-01; First posted 2017-10-04 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Beliefs; Disability Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retrain pain educational website (Experimental): Participants will be invited to consult an educational website developped for patients with chronic pain
  Interventions: Other: Retrain pain educational website
- Booklet (Experimental): Participants will be invited to read an educational booklet for patients with chronic pain
  Interventions: Other: Booklet
- Control (No Intervention): Participants in this group will receive the 2 educational tools at the end of the study

INTERVENTIONS:
Other: Retrain pain educational website — Patients in this group will be invited to consult an educational website developped for patients with chronic pain
  Arms: Retrain pain educational website
Other: Booklet — Patients in this group will be invited toread an educational booklet developped for patients with chronic pain
  Arms: Booklet

SUMMARY:
This trial aims at comparing the effectiveness of different didactic tools developed for patients with chronic pain to correct misbeliefs and improve disability in patients with chronic low back pain

DETAILED DESCRIPTION:
This trial aims at comparing the effectiveness of different didactic tools (an educational website vs a booklet) developed for patients with chronic pain to correct misbeliefs and improve disability in patients with chronic low back pain.

Participants of the 2 experimental groups will be invited to use the tool they receive during a one-month period.

ELIGIBILITY:
Inclusion Criteria:

* individuals with non-specific persistent low back pain (pain > 6 months) who had their pain assessed by their general practitioner or a specialist within the last 3 months

Exclusion Criteria:

* specific low back pain,
* educational treatment (back school, cognitive-behavioral, pain neurosciences education) in progress or planned during the study period
* previous consultation of the didactic tools investigated in the present study
* nerve root compromise,
* recent spinal surgery (<3 months)
* not fluent in French
* no regular access to a computer and the internet
* present follow-up by a psychiatrist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire | Change from baseline to the three-month follow-up
  Questionnaires to test patients' beliefs
Roland-Morris Disability Questionnaire | Change from baseline to the three-month follow-up
  Disability questionnaire

SECONDARY OUTCOMES:
Brief-Illness Perception Questionnaire | Baseline, one month after receiving the tool, one-month follow-up and three-month follow-up
  Questionnaire about patients' beliefs/representations
Back-PAQ questionnaire | Baseline, one month after receiving the tool, one-month follow-up and three-month follow-up
  Questionnaire about patients' beliefs
Pain intensity | Baseline, one month after receiving the tool, one-month follow-up and three-month follow-up
  Pain Numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Demoulin, Principal Investigator — Liege University Hospital
Locations (1):
- Liege University Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No